CLINICAL TRIAL: NCT01102387
Title: Phase IIa, Two-centre, Randomized, Double Blind Study to Evaluate the Anti-mycotic and Anti-inflammatory Efficacy of Topical Combinational Product LAS41003 Versus Corresponding Mono-substances in Patients With Candida Infections in Intertriginous Areas at the Trunk
Brief Title: Efficacy and Safety of LAS41003 in the Treatment of Intertriginous Candida Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H 552 000 - 0920; 2009-016627-56 (EudraCT Number)
Record Dates: First submitted 2010-03-30; First posted 2010-04-13 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2011-01

CONDITIONS: Candidiasis
Keywords: Candida infections in intertriginous areas
MeSH Terms: conditions — Candidiasis | interventions — octenidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LAS41003 (Experimental)
  Interventions: Drug: LAS41003
- LAS189962 (Active Comparator)
  Interventions: Drug: LAS189962
- LAS189961 (Active Comparator)
  Interventions: Drug: LAS189961

INTERVENTIONS:
Drug: LAS41003 — Once daily, topically
  Arms: LAS41003
Drug: LAS189962 — Once daily, topically
  Arms: LAS189962
Drug: LAS189961 — Once daily, topically
  Arms: LAS189961

SUMMARY:
The aim of this study is to determine the efficacy and safety of once daily topical application of the combinational cream LAS41003 compared to the corresponding mono-substances in the treatment of candida infections in intertriginous areas at the trunk.

ELIGIBILITY:
Inclusion Criteria:

* presence of candida infections in one or more intertriginous areas (trunk), confirmed by positive mycological sample at baseline;
* female volunteers of childbearing potential must either be surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of less than 1 % per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra uterine devices [IUDs], sexual abstinence or vasectomized partner;
* written informed consent

Exclusion Criteria:

* receiving systemic therapy with cytotoxic or immunosuppressive drugs either concurrently or within 12 weeks before the baseline visit;
* patients who have been treated with oral anti-fungal agents within the 12 weeks prior to study entry or treated with topical anti-fungal agents on the intertrigines within the previous 2 weeks;
* evidence of drug or alcohol abuse;
* pregnancy or nursing;
* symptoms of a clinically significant illness that may influence the outcome of the study in the four weeks before and during the study;
* treatment with any other investigational drug in the four weeks preceding the study;
* known allergic reactions to components of the study preparations, hypersensitivity against cetylstearyl alcohol;
* treatment with systemic or locally acting medications which might counter or influence the study aim within two weeks before the beginning of the study (e.g. glucocorticosteroids);
* in the opinion of the investigator or physician performing the initial examination the subject should not participate in the study, e.g. due to probable non-compliance or inability to

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy and mycological culture | Day 14
  Clinical assesment scores and mycological status of candida (mycological culture)

SECONDARY OUTCOMES:
Physical examination, AEs | 14 Days
  Physician assesmentes of sign and symptoms (erythema, papules, pustules and maceration)
  Percentage of local skin reactions, AEs

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Willers, MD, MBA, Study Director — Almirall Hermal GmbH
Locations (6):
- Germany (6):
  - Investigational Site #5, Augsburg
  - Investigational Site #4, Bad Saarow
  - Investigational Site #2, Berlin
  - Investigational Site #6, Dülmen
  - Investigational Site #1, Hamburg
  - Investigational Site #3, Vechta

REFERENCES:
- See also: Almirall Corporate Website — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp